CLINICAL TRIAL: NCT05377138
Title: Evaluate and Optimize a Virtual Care Model for PrEP Delivery: Pilot Study
Brief Title: Evaluate and Optimize an Online Care Model for PrEP Delivery: Pilot Study
Acronym: ePrEP Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Fred Hutchinson Cancer Center (Other); Jomo Kenyatta University of Agriculture and Technology (Other); Partners in Health & Research Development (Unknown); MYDAWA (Unknown); Audere (Unknown)
Responsible Party: Principal Investigator, Monisha Sharma, Assistant Professor, School of Public Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00014987
Record Dates: First submitted 2022-04-19; First posted 2022-05-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: Online PrEP; PEP; Online PEP; pharmacies; HIV prevention; Kenya
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: MYDAWA clients determined to be eligible for PrEP or PEP following online screening and a remote meeting with a MYDAWA clinical officer will be delivered a blood-based HIV self-test followed by daily oral PrEP or PEP) at home and continued remote HIV prevention (i.e., PrEP) support for a small fee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MYDAWA clients (Experimental): MYDAWA clients determined to be eligible for PrEP or PEP can order them online and have them delivered a small fee. This is not currently the standard of care in Kenya. Those who are not in the study can only receive PrEP or PEP at healthcare facilities in Kenya.
  Interventions: Other: Online PEP/PrEP delivery

INTERVENTIONS:
Other: Online PEP/PrEP delivery — Delivery of PEP or PrEP after online consultation and HIVST image upload.

SUMMARY:
Daily oral pre-exposure prophylaxis (PrEP) is highly effective at preventing HIV acquisition, but uptake in Kenya remains low. Barriers to clinic-based PrEP delivery exist (e.g., long wait times, stigma), thus the delivery of PrEP via online pharmacy platforms has the potential to expand the reach of PrEP access in Kenya. In this pilot study, the investigators will test a new model of PrEP delivery that has never been tried in a sub-Saharan African setting: online pharmacy-delivered PrEP. The investigators will work in collaboration with MYDAWA, an online pharmacy in Kenya, to deliver PrEP on their platform for 18 months. Online PrEP delivery will include a PrEP eligibility assessment, HIV self-test delivery, a remote clinical encounter, PrEP medication delivery, and virtual PrEP support tools. If a participant is identified as eligible for pre-exposure prophylaxis (PEP), then PEP will be prescribed for 29 days and the participant will be asked to make another appointment at the end of this time to reassess for PrEP eligibility. The investigators will measure PrEP uptake and continuation over time and also measure a number of implementation outcomes, including acceptability and costs. The investigators anticipate that online pharmacy PrEP delivery will result in high uptake and continuation (similar to that or greater than public clinics), will be acceptable to clients, and will be low cost.

DETAILED DESCRIPTION:
Online PrEP may help overcome patient- and provider-level barriers to facility-delivered PrEP. At the patient-level, online PrEP may increase privacy and convenience by enabling patients to receive PrEP at a location and time of their choice. Additionally, by expanding options for PrEP delivery, patients can select a model that fits their preferences. The delivery of PrEP directly via couriers may also decrease the time patients spend (and costs associated with) traveling to and waiting at health facilities, and the stigma associated with visiting HIV clinics for PrEP care. At the provider-level, online PrEP may decrease crowding at facilities and increase the time providers can spend with patients seeking treatment services. Additionally, shifting some PrEP delivery responsibilities to lower-paid couriers may be cost saving to the health system. Together, these advantages of online PrEP may increase PrEP continuation among individuals at risk for HIV.

MYDAWA, Kenya's first licensed online pharmacy (https://mydawa.com), is uniquely positioned to support online PrEP delivery by applying technology to deliver essential medicines and health supplies to local communities.

The overall goal of this study is to generate data to support the relevant policy decisions regarding broader adoption of online PrEP delivery in the region. The investigators plan to develop and evaluate the feasibility of a online delivery model to support PrEP initiation and continuation among individuals at risk of HIV acquisition in Kenya. The model will deliver once-daily oral tenofovir/emtricitabine (TDF/FTC). To evaluate the feasibility of this model in Kenya, the investigators propose testing the uptake of a "minimally viable" model, understanding the characteristics of online PrEP clients and the acceptability of the model among these clients, and evaluating the costs associated with the model.

Specific objectives

1. To develop and pilot test a model of online PrEP delivery on PrEP initiation and continuation outcomes among individuals at risk of HIV acquisition in Kenya.
2. To evaluate the acceptability, appropriateness, feasibility, and costs of an online PrEP delivery model in Kenya.

Hypothesis The investigators hypothesize that an online PrEP delivery model will address patient- and provider-level barriers to clinic-delivered PrEP and result in high PrEP initiation and continuation (compared to facility-based models), be acceptable and appropriate and providers and clients, and low-cost.

ELIGIBILITY:
Inclusion criteria:

* Accessed MYDAWA Services for HIVST or requested PrEP information through MYDAWA
* Are interested in and willing to take PrEP and are willing to pay for the PrEP delivery cost
* Be willing to pay for a blood-based HIVST and delivery cost
* Self-reported HIV negative
* Are able to access the MyDAWA platform using computer or a smartphone for the duration of the study
* Are able to access the internet
* Are able to read and comprehend English
* Are living in or willing to travel to the Nairobi area to receive virtual PrEP services
* Are able and willing to provide informed consent electronically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2357 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
PrEP initiation | 1 year
  % of participants that were delivered PrEP among those screened for HIV risk and determined PrEP eligible via the online (MYDAWA) platform.
PrEP continuation: refills with 45 days of PrEP initiation | 1 year
  % of participants who refilled PrEP within 45 days of first PrEP delivery among those screened for HIV risk and determined PrEP eligible via the online (MYDAWA) platform.
PEP initiation | 1 year
  % of participants that were delivered PEP among those screened for HIV risk and determined PEP eligible via the online (MYDAWA) platform.

SECONDARY OUTCOMES:
PrEP continuation: any refills | 1 year
  % of participants who refilled PrEP (at least once) among those screened for HIV risk and determined PrEP eligible via the online (MYDAWA) platform.
PrEP continuation => 2 refills | 1 year
  % of participants who refilled PrEP (at least twice) among those screened for HIV risk and determined PrEP eligible via the online (MYDAWA) platform.
PrEP stopping and restarting | 1 year
  % of participants who refilled PrEP (at least once) with a gap of at least 14 days between when their pills would runt out and the next delivery of pills, among those screened for HIV risk and determined PrEP eligible via the online (MYDAWA) platform.
PrEP pill coverage | 1 year
  % of PrEP pill coverage among days at HIV risk among clients that initiated PrEP
Self-reported PrEP use/adherence | 1 year
  Self-reported PrEP use/adherence
Transition from PEP to PrEP | 1 year
  % of clients that initiated PrEP among those what received PEP via MYDAWA
Feasibility of implementing online PrEP | 1 year
  To what extent can online PrEP be successfully delivered to intended participants in the Kenyan context?
Acceptability of online PrEP | 1 year
  To what extent is online PrEP judged as suitable, satisfying, or attractive to clients?
Cost associated with online PEP delivery | 1 year
  Cost to deliver PEP to each PEP client
Cost associated with online PrEP delivery | 1 year
  Cost per client month on PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Monisha Sharma, PhD, MSPH, Principal Investigator — University of Washington; Katrina F Ortblad, ScD, MPH, Principal Investigator — Fred Hutch Cancer Center
Locations (1):
- Jomo Kenyatta University of Agriculture and Technology, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No